CLINICAL TRIAL: NCT03600454
Title: The Effect of Anesthesia on Perioperative Muscle Weakness and Neuro-endocrine Stress Response
Acronym: MUSCLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Dimitri Dylst, Principal Investigator, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 18/0010U
Record Dates: First submitted 2018-06-14; First posted 2018-07-26 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Muscle Weakness; Anesthesia; Anesthesia, Local; Surgery
MeSH Terms: conditions — Muscle Weakness | interventions — Anesthesia, General; Anesthesia, Spinal; Analgesia, Epidural

STUDY DESIGN:
Intervention Model Description: Two independent, but complimentary, studies will be performed to evaluate the primary objective and the secondary objectives in this prospective trail.
  Group 1: The effect of spinal anesthesia as compared to general anesthesia for total hip arthroplasty
  Group 2: The effect of epidural analgesia compared to general anesthesia alone for major abdominal surgery
Who Masked: Investigator
Masking Description: Patients will be randomized using a computer-generated permuted block randomization sequence (variable block-size, 1:1 allocation). The randomization will be determined on the preoperative anesthesia assessment. After the randomisation, the investigator will inform the patient which anesthesia he/she will get during the operation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Hip surgery: spinal anesthesia (Experimental): Patients scheduled to undergo elective total hip arthroplasty will receive spinal anesthesia in combination with monitored anesthesia care (MAC).
  Interventions: Drug: Spinal anesthesia
- Hip surgery: general anesthesia (Experimental): Patients scheduled to undergo elective total hip arthroplasty will receive general anesthesia
  Interventions: Drug: General anesthesia
- Colectomy: general anesthesia and epidural analgesia (Experimental): Patients scheduled to undergo elective laparoscopic hemicolectomy will receive general anesthesia combined with epidural analgesia (EA).
  Interventions: Drug: General anesthesia and epidural analgesia
- Colectomy: general anesthesia (Experimental): Patients will receive general anesthesia.
  Interventions: Drug: General anesthesia

INTERVENTIONS:
Drug: General anesthesia — The induction of general anesthesia will be delivered in a standardized manner with the intravenous administration of fentanyl 2µg/kg and propofol
  Arms: Colectomy: general anesthesia; Hip surgery: general anesthesia
Drug: Spinal anesthesia — The level of puncture will be L4 - L5. 10 mg bupivacaine will be injected in the subarachnoid space, after spontaneous surge of cerebrospinal fluid
  Arms: Hip surgery: spinal anesthesia
Drug: General anesthesia and epidural analgesia — The induction of general anesthesia will be delivered in a standardized manner with the intravenous administration of fentanyl 2 µg/kg and propofol. A thoracic epidural catheter will be placed with 3 ml of xylocaine 2% (with epinephrine 1/200.000).
  Arms: Colectomy: general anesthesia and epidural analgesia

SUMMARY:
The effect of surgery, in contrary to critical illness, on muscle weakness hasn't been thoroughly investigated. Recent data suggest that elective surgery may also induce muscle weakness. The neuro-endocrine stress response could be involved in the pathophysiology. Whether the mode of anesthesia/analgesia can influence muscle weakness, by influencing the neuro-endocrine stress response is unknown. Gaining insight in this matter could affect quality of care and benefit patient recovery and satisfaction.

DETAILED DESCRIPTION:
In this study, the investigators want to demonstrate whether the application of neuraxial anesthesia for elective surgery diminishes perioperative muscle weakness. Since spinal and epidural anesthesia/analgesia have been shown to influence the neuro-endocrine stress response, the possible underlying mediator of perioperative muscle weakness, the investigators will perform two different, but complementary, studies. In one study, patients scheduled for elective total hip arthroplasty will receive spinal anesthesia, without losing consciousness and maintaining a free airway, as compared to receiving general anesthesia. In another study, patients scheduled for a laparoscopic hemicolectomy will receive epidural anesthesia/analgesia during and after the surgery as compared to receiving no epidural anesthesia/analgesia. These studies allow the investigators to identify whether the application of neuraxial anesthesia/analgesia could diminish perioperative weakness and allow us to identify other possible mediators of perioperative muscle weakness, such as losing consciousness or receiving neuromuscular blockade.

This study has the potential to help to identify a new side-effect of elective surgery, namely perioperative muscle weakness, and to identify a possible treatment for this possible new complication, namely neuraxial anesthesia and analgesia, which might benefit many patients in the future. Furthermore, investigating the possible mediating role of the neuro-endocrine stress response might identify new therapeutic targets, such as glucagon modulation.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older.
* Scheduled for elective total hip arthroplasty or hemicolectomy.

Exclusion Criteria:

* Lack of informed consent or inability to give informed consent.
* Urgent surgery, such as hip fracture.
* Contra-indications for spinal or epidural analgesia, including but not limited to:

  * Infection at the site of puncture.
  * Coagulopathy.
  * Severe hypovolemia.
  * Severe aortic valve stenosis (cross sectional area < 1,3 cm2).
  * Severe mitralis valve stenosis (cross sectional area < 1,0 cm2).
  * Increased intracranial pressure.
  * Pre-existing neurological condition.
  * Severe spine deformity.
  * Sepsis.
  * Body mass index (BMI) > 35 kg/m2
* Hypersensitivity or known allergic reactions to any products used for anesthesia.
* History of chronic opioid analgesics use.
* Preoperative use of steroids:

  * Including, but not limited to: injection of hydrocortisone < 3 months before surgery.
* Preexisting muscle disease

  * Including, but not limited to: Steinert's disease, amyotrophic lateral sclerosis (ALS), Duchenne dystrophy, amputation of dominant arm or hand.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-18 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in post-operative peripheral limb muscle weakness | Pre-operative (Day 0) and postoperatively (Day 1, Day 7 and Day 28)
  The strength will be measured in the dominant hand using a Camry handgrip Dynamometer. The measurement will take place on the first day postoperatively, at day 7 and day 28 and will be compared to the preoperative measurement during the preoperative assessment

SECONDARY OUTCOMES:
Change in general health status | Pre-operative (Day 0) and postoperatively (Day1, Day7 and Day28)
  Measuring generic health status by the EQ-5D questionnaire preoperatively and at day 1, 7 and 28 after surgery. The general health status is scored by severity ranging from 0 (no problems) to 5 (severe problems)
Change in post-operative lung function: vital capacity | Pre-operative (Day 0) and postoperatively (Day 1, Day 7 and Day 28)
  Post-operative lung function at day 1, 7 and 28. The investigators will measure vital capacity (VC). These measurements will take place preoperatively and day 1, 7 and 28 after surgery, using a portable pulmonary function testing machine (PPFTM).
Change in post-operative lung function:forced expiratory volume | Pre-operative (Day 0) and postoperatively (Day 1, Day 7 and Day 28)
  Post-operative lung function at day 1, 7 and 28. The investigators will measure forced expiratory volume in 1 second (FEV1). These measurements will take place preoperatively and day 1, 7 and 28 after surgery, using a portable pulmonary function testing machine (PPFTM).
Change in the neuro-endocrine stress response: Cortisol | Pre-operative (Day 0), end of surgery and postoperatively (Day 1)
  Blood samples will be taken at the start, end of surgery and the day after surgery to measure cortisol (nmol/L) in the samples
Change in the neuro-endocrine stress response: ACTH | Pre-operative (Day 0), end of surgery and postoperatively (Day 1)
  Blood samples will be taken at the start, end of surgery and the day after surgery to measure ACTH (nmol/L) in the samples
Change in the neuro-endocrine stress response: Noradrenaline | Pre-operative (Day 0), end of surgery and postoperatively (Day 1)
  Blood samples will be taken at the start, end of surgery and the day after surgery to measure noradrenaline (nmol/L) in the samples
Change in glycemia levels | Pre-operative (Day 0), end of surgery and postoperatively (Day 1)
  Measurement of glycemia in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitri Dylst, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

REFERENCES:
- [Derived] Van Boxstael S, Peene L, Dylst D, Penders J, Hadzic A, Meex I, Corten K, Mesotten D, Thiessen S. The effect of spinal versus general anaesthesia on perioperative muscle weakness in patients having bilateral total hip arthroplasty: a single center randomized clinical trial. Eur J Med Res. 2023 Oct 20;28(1):450. doi: 10.1186/s40001-023-01435-6. PMID 37864209